CLINICAL TRIAL: NCT06865404
Title: Additive Regional Fascial Plain Blocks to Pectointercostal Fascial Block for Postoperative Pain Management After Cardiac Surgery: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRP 00012098
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain Management
Keywords: pain; sternotomy; cardiac surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pecto-Intercostal Fascial Plane Block technique (Experimental): The ultrasound probe will be positioned parallel and 2-3 cm lateral from the midline in the 4th or 5th intercostal space. The needle will be inserted in-plane in a cauda-cranial direction until the tip of the needle reaches the plane of the fascia between the pectoralis major muscle and the external intercostal muscles. A 20 ml volume of bupivacaine 0.25% will be injected on each side.
  Interventions: Procedure: PIFPB block
- Pecto-Intercostal Rectus Sheath Fascial Plane Block technique (14) (Active Comparator): After the PIFPB is performed with the same position and probe, a bilateral posterior rectus sheath block (PRSB) will be conducted. The probe will be placed 2-3 cm next to the xiphoid in the epigastric region and parallel to the costal margin. The needle will be inserted into the plane between the rectus abdominal muscle and its posterior sheath. After verifying needle placement, 10 ml of bupivacaine 0.25% will be injected on each side.
  Interventions: Procedure: PIRSB Block
- Pecto-intercostal facial plane with an external oblique intercostal block (Active Comparator): After the PIFPB is performed with the same position and probe, an external oblique block will be used to place the linear array ultrasound probe between the midclavicular line and the anterior axillary line at the level of the 6th rib, with the direction mark pointing to the cephalad. The probe will be rotated on the slightly medial cranial end, and the caudal end will be lateral to produce a mesial sagittal oblique view and a short-axis view of the ribs. The following structures will be identified from superficial to deep layers: subcutaneous tissue, external oblique muscle, intercostal muscles, pleura, and lung. After determining the thoracic fascial space between the external oblique muscle and the intercostal muscles, bupivacaine 20 mL will be slowly injected into the space with a nerve block needle at the head side of the 6th rib horizontally near the mid axillary line. The block will be repeated

INTERVENTIONS:
Procedure: PIFPB block — The ultrasound probe will be positioned parallel and 2-3 cm lateral from the midline in the 4th or 5th intercostal space. The needle will be inserted in-plane in a cauda-cranial direction until the tip of the needle reaches the plane of the fascia between the pectoralis major muscle and the external intercostal muscles. A 20 ml volume of bupivacaine 0.25% will be injected on each side.
  Arms: Pecto-Intercostal Fascial Plane Block technique
Procedure: PIRSB Block — After the PIFPB is performed with the same position and probe, a bilateral posterior rectus sheath block (PRSB) will be conducted. The probe will be placed 2-3 cm next to the xiphoid in the epigastric region and parallel to the costal margin. The needle will be inserted into the plane between the rectus abdominal muscle and its posterior sheath. After verifying needle placement, 10 ml of bupivacaine 0.25% will be injected on each side.
  Arms: Pecto-Intercostal Rectus Sheath Fascial Plane Block technique (14)
Procedure: PIEOB block — After the PIFPB is performed with the same position and probe, an external oblique block will be used to place the linear array ultrasound probe between the midclavicular line and the anterior axillary line at the level of the 6th rib, with the direction mark pointing to the cephalad. The probe will be rotated on the slightly medial cranial end, and the caudal end will be lateral to produce a mesial sagittal oblique view and a short-axis view of the ribs. The following structures will be identified from superficial to deep layers: subcutaneous tissue, external oblique muscle, intercostal muscles, pleura, and lung. After determining the thoracic fascial space between the external oblique muscle and the intercostal muscles, bupivacaine 20 mL will be slowly injected into the space with a nerve block needle at the head side of the 6th rib horizontally near the mid axillary line. The block will be repeated in the same way on the other side.

SUMMARY:
Acute postoperative pain is severe in cardiac patients undergoing sternotomy, and pain intensity is more severe than expected. Many patients referred to tube insertion as the most painful site after coronary artery bypass surgery. (6) Rectus sheath block (RSB) can offer somatic analgesia for midline incisions. (7) It has been verified to manage subxiphoid drainage pain effectively and safely for cardiac surgery patients. Another intervention, External oblique intercoastal plane block (EOIPB) is given at the mid-clavicular line and may block the intercostal nerve's anterior and lateral branches. Anesthesia is provided between the external oblique and intercostal nerves. This allows analgesia of the anterior upper abdominal wall between T6-T10 dermatomes in the anterior axillary line and T6-T9 dermatomes in the midline. It blocks the lateral and anterior branches of T6-T10 intercostal nerves.

DETAILED DESCRIPTION:
Additive regional fascial plain blocks to pectointercostal fascial block for postoperative pain management after cardiac surgery: a randomized controlled trial

Introduction Acute postoperative pain is severe in cardiac patients undergoing sternotomy, and pain intensity is more severe than expected. (1) Poorly controlled pain after surgery can lead to myocardial ischemia and pulmonary infections. (2) A perioperative multimodal opioid-sparing pain management plan is recommended to accelerate recovery. (3) Novel fascial regional techniques such as pectointercostal fascial block (PIFB) have been applied in cardiac surgery and have achieved satisfying analgesia. (4, 5) However, postoperative pain in cardiac surgery is a multidimensional phenomenon that involves incision, sternal retraction, musculoskeletal trauma, and drainage catheter insertion sites. Many patients referred to tube insertion as the most painful site after coronary artery bypass surgery. (6) Rectus sheath block (RSB) can offer somatic analgesia for midline incisions. (7) It has been verified to manage subxiphoid drainage pain effectively and safely for cardiac surgery patients. (8) Fascial plane blocks in regional anesthesia have gained importance in recent years. It involves injection into a tissue plane to provide analgesia and is an alternative to neuraxial and paravertebral techniques. It is often safer and is associated with less cardiorespiratory instability or complications compared to epidural analgesia (9). External oblique intercoastal plane block (EOIPB) is given at the mid-clavicular line and may block the intercostal nerve's anterior and lateral branches. Anesthesia is provided between the external oblique and intercostal nerves. This allows analgesia of the anterior upper abdominal wall between T6-T10 dermatomes in the anterior axillary line and T6-T9 dermatomes in the midline. It blocks the lateral and anterior branches of T6-T10 intercostal nerves. (10) With a considerable incidence of epigastric drain site pain reported after the pectointercostal fascial plane block, we will conduct this clinical trial to find an additive regional block.

Objectives The primary objective of the study is to report the incidence of non-sternal epigastric drain site pain after ultrasound-guided bilateral pectointercostal fascial plane block (PIFPB), a pectointercostal facial plane with posterior rectus sheath plane block (PIPRSB), and pectointercostal facial plain with external oblique for acute postoperative pain after sternotomy in adult cardiac surgery patients. The secondary objectives will include intravenous opioid consumption 24 hours after ICU admission, time to extubation, the intensity of postoperative pain, time to 1st rescue analgesia, patient satisfaction, and any possible side effects of the study drugs and technique.

Methodology A double-blind, randomized control trial will be conducted after approval from the institutional ethical committee, and the trial will be registered with the clinical trial registry. The trial will be conducted at Alexandra University Hospital. The selection of patients will be based on inclusion criteria. The study will comply with the principles outlined in the Declaration of Helsinki. After explaining the nature and purpose of the trial, informed consent will be obtained from all participants. Before enrolling the patients, the procedure will be described, and informed consent will be taken for making facial plain blocks in the three groups.

Inclusion Criteria: The study will include adult patients of both sexes aged 18 to 60 who are scheduled to have fast-tracking elective on-pump cardiac surgery through a median sternotomy with epigastric drain insertion.

Exclusion Criteria: patients who refused to participate in the study, also who had Cognitive impairment or mental disorders, Ages <20 and >65 years, BMI <18 and >35, patients with puncture site infection, patients who documented allergy to local anesthetic drugs, patients used to take chronic pain medications, patients who made previous sternotomy or chest surgery and patients with a history of substance abuse.

After assessing the inclusion criteria, 150 patients will be randomized using a computer-generated randomization sequence. These selected patients will be divided into three groups. Group allocation will be done using a sealed envelope technique, and patients will be allocated equally to the three groups.

Groups:

PIFPB Group: Participants will receive ultrasound-guided Pecto-intercostal fascial plane block.

PIRSB Group: Participants will receive an ultrasound-guided Pectointercostal-posterior rectus sheath plane block.

PIEOB Group: Participants will receive an ultrasound-guided Pectointercostal facial plane with an external oblique block

Methods:

Preoperative evaluation Participants will be subjected to history taking, complete physical examinations, laboratory investigations, a chest X-ray, standard 12 leads electrocardiogram, echocardiogram, and other investigations as needed at admission. All Patients will be informed about the technique of each block, and written consent will be obtained from every patient. Each patient will be taught to use the numerical rating scale (NRS) to measure pain intensity. (11) Anaesthesia Technique

Monitoring:

Electrocardiography (ECG), invasive arterial blood pressure (IABP) in mmHg, central venous pressure (CVP) in mmHg, peripheral oxygen saturation percentage (SpO2%), end-tidal carbon dioxide tension (EtCO2) in mmHg, core temperature using nasopharyngeal temperature probe (°C), urine output (ml/hour), arterial blood gases, activated clotting time (ACT) will be continuously monitored during the whole procedure.

Cannulation:

On arrival at the operating theatre, the patients will receive oxygen via face mask (6 L/min). Cannulation will be done with a peripheral large bore (16-18 G) intravenous catheter under local anesthesia. Mild sedation with intravenous midazolam and fentanyl will be done. An arterial line catheter will be inserted using a local anesthetic to monitor arterial pressure. After anesthesia induction, central venous cannulation of the right internal jugular will be performed under ultrasound guidance.

Induction:

For induction of anesthesia, midazolam (0.05-0.1 mg/kg), fentanyl (2-5 mg/kg), propofol (1-2 mg/kg), and rocuronium (1 mg/kg) will be administered intravenously (IV). Mechanical ventilation will be started after tracheal intubation with a suitable-sized cuffed oral endotracheal.

Maintenance:

To maintain anesthesia while maintaining hemodynamic parameters (20% of baseline for heart rate and blood pressure), inhalation of isoflurane (MAC 1%-2%), an air-oxygen mixture, IV rocuronium boluses (0.6 mg/kg), and if necessary, IV fentanyl (1 µg /kg) boluses will be used.

Surgical approach:

Median sternotomy and cardiopulmonary bypass will be used. For all patients, per the hospital's practice, drains will be placed through separate stab incisions after cardiac procedures, typically near the inferior aspect of the sternotomy incision (epigastric region). One or two drains were placed anteriorly, overlying the heart (retrosternal epigastric drain). If either pleural space were opened during the procedure, a drain would be put into the dependent portion of the pleural space through an epigastric incision (pleural space epigastric drain). It will be removed mainly by the third postoperative day after surgical consultation.

Regional fascial plan blocks procedures:

Immediately after surgery, with the patient in the supine position, bilateral ultrasound-guided fascial plan blocks will be done in the operating room. A linear-array ultrasound transducer probe guided the in-plane needle approach at high frequencies (8-13 MHz). A block needle (80- -mm long, 22-gauge short bevel; Stimuplex Ultra 360, B. Braun, Germany) will be advanced from caudal to cranial until the needle end is in the desired plane, with aseptic measures always taken. The separation of the fascial layers during a test bolus (1-2 mL) of normal saline administered (in real-time) confirmed the needle's precise placement. On each side, after excluding intravascular and intrapleural puncture, the volume of 0.25% bupivacaine (12) will be injected into the fascial plane at a maximum dose of 2.5 mg/kg. At the same time, real-time imaging for the fascial plane's separation and the local anesthetic (LA) spread was performed during the injection. The patient will be attentively monitored for 30 minutes after the block is completed for signs of toxicity, hemodynamic instability, and allergic reactions.

Pecto-Intercostal Fascial Plane Block technique (13) The ultrasound probe will be positioned parallel and 2-3 cm lateral from the midline in the 4th or 5th intercostal space. The needle will be inserted in-plane in a cauda-cranial direction until the tip of the needle reaches the plane of the fascia between the pectoralis major muscle and the external intercostal muscles. A 20 ml volume of bupivacaine 0.25% will be injected on each side.

Pecto-Intercostal Rectus Sheath Fascial Plane Block technique (14) After the PIFPB is performed with the same position and probe, a bilateral posterior rectus sheath block (PRSB) will be conducted. The probe will be placed 2-3 cm next to the xiphoid in the epigastric region and parallel to the costal margin. The needle will be inserted into the plane between the rectus abdominal muscle and its posterior sheath. After verifying needle placement, 10 ml of bupivacaine 0.25% will be injected on each side.

Pecto-intercostal facial plane with an external oblique intercostal block (10, 15) After the PIFPB is performed with the same position and probe, an external oblique block will be used to place the linear array ultrasound probe between the midclavicular line and the anterior axillary line at the level of the 6th rib, with the direction mark pointing to the cephalad. The probe will be rotated on the slightly medial cranial end, and the caudal end will be lateral to produce a mesial sagittal oblique view and a short-axis view of the ribs. The following structures will be identified from superficial to deep layers: subcutaneous tissue, external oblique muscle, intercostal muscles, pleura, and lung. After determining the thoracic fascial space between the external oblique muscle and the intercostal muscles, bupivacaine 20 mL will be slowly injected into the space with a nerve block needle at the head side of the 6th rib horizontally near the mid axillary line. The block will be repeated in the same way on the other side.

Postoperative care:

All anesthetics will be discontinued after surgery, and patients will be transferred to the intensive care unit, where they will be mechanically ventilated under monitoring for extubation and further medical care. Per the standard ICU policy, patients will be extubated as soon as it is clinically feasible after surgery. Participants received paracetamol IV (1 g every 8 hours) and fentanyl infusion (1 µg/kg/h) intravenously starting at the end of the surgery and will continue in the ICU until extubation. After extubation, participants will be instructed to ask for analgesia if their NRS score at rest is >4. On the patient's request, one µg/kg of intravenous fentanyl will be administered after extubation when the NRS is > four at rest. If the patient's pain persists after two fentanyl doses administered over 60 minutes, a 1-µg/kg/h fentanyl infusion will be started

Measurements:

1. Demographic and baseline data: Age (years), sex, weight (Kg), BMI (kg/m2), physical status (ASA scores), type of surgical procedure, aortic cross-clamping time (min), cardiopulmonary bypass time (min), total duration of surgery (min), and total dose of fentanyl (µg/kg) administered intraoperatively will be recorded.
2. Indicine of non-sternal wound pain: Ask the patients about the site of pain. Is it at the sternal wound or the epigastric drain?
3. Postoperative opioid consumption: total dose of fentanyl (µg/kg) administered postoperatively during the first postoperative 24 h after ICU admission.
4. Time to extubation: duration (minutes) between ICU admission and endotracheal extubation.
5. Pain Assessment: NRS score (0-10) will be assessed at rest and cough. It will be measured immediately after extubation and 2, 4, 8, 12, and 24 hours after ICU admission.
6. Time of first rescue analgesia: time (minutes) until the first request of fentanyl analgesia will be recorded from ICU admission time.
7. Incidence of adverse:

   1. Related to local anesthesia toxicity (neurologic or cardiovascular events).
   2. Related to block procedure (hematoma and pneumothorax).
   3. Related to opioid administration (postoperative nausea and vomiting, dizziness, and pruritus).

Data Collection: Data will be collected by trained research personnel, entered into a secure database, and maintained following Good Clinical Practice (GCP) guidelines.

Data Analysis: Statistical analysis will be performed using appropriate tests to compare primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

The study will include adult patients of both sexes aged 18 to 60 who are scheduled to have fast-tracking elective on-pump cardiac surgery through a median sternotomy with epigastric drain insertion.

Exclusion Criteria:

* patients who refused to participate in the study, also
* who had Cognitive impairment or mental disorders,
* Ages <20 and >65 years,
* BMI <18 and >35,
* patients with puncture site infection,
* patients who documented allergy to local anesthetic drugs,
* patients used to take chronic pain medications,
* patients who made previous sternotomy or chest surgery and
* patients with a history of substance abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
To compare the incidence of non-sternal epigastric drain site pain after ultrasound-guided bilateral PIFPB, PIPRSB, and PIEOB for acute postoperative pain after sternotomy in adult cardiac surgery patients | 24 hours postoperatively
  Incidence of non-sternal wound pain by asking the patients about the site of pain. Is it at the sternal wound or the epigastric drain?

SECONDARY OUTCOMES:
Recording intravenous opioid consumption 24 hours after ICU admission | 24 hours postoperatively
  total dose of fentanyl (µg/kg) administered postoperatively is recorded.
Time to extubation | 24 hours postoperatively
  It is the duration (minutes) between ICU admission and endotracheal extubation.
the intensity of postoperative pain & time to 1st rescue analgesia | 24 hours postoperatively
  Pain Assessment using NRS score (0-10) will be assessed at rest and cough. It will be measured immediately after extubation and 2, 4, 8, 12, and 24 hours after ICU admission.
  Time of first rescue analgesia: time (minutes) until the first request of fentanyl analgesia will be recorded from ICU admission time.
possible side effects of the study drugs and technique. | 24 hours postoperatively
  Incidence of adverse:
  1. Related to local anesthesia toxicity (neurologic or cardiovascular events).
  2. Related to block procedure (hematoma and pneumothorax).
  3. Related to opioid administration (postoperative nausea and vomiting, dizziness, and pruritus).

CONTACTS AND LOCATIONS:
Overall Officials: Islam Elbardan, Dr, Principal Investigator — University of Alexandria
Locations (1):
- Alexandria University, Alexandria, Alexandria Governorate, Egypt